CLINICAL TRIAL: NCT00320983
Title: A Phase I Study of Adjuvant Topotecan and Cisplatin With Concurrent Radiation Therapy for Advanced Cervical Cancer
Brief Title: Study of Adjuvant Topotecan and Cisplatin With Concurrent Radiation Therapy for Advanced Cervical Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Harriet O Smith, MD; Principal Investigator, University of New Mexico CRTC
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1601C
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2008-10

CONDITIONS: Cervical Cancer
Keywords: Cancer; Cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms | interventions — Topotecan; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Topotecan — Topotecan
  Other Names: Hycamtin
Drug: Cisplatin — Cisplatin
  Other Names: Platinol AQ

SUMMARY:
A Phase I Study of Adjuvant Topotecan and Cisplatin with Concurrent Radiation Therapy for Advanced Cervical Cancer.

DETAILED DESCRIPTION:
Examines the effects of Topotecan and Cisplatin with radiation for advanced cervical cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed advanced cervical carcinoma who, following optional surgical staging, are not deemed to be curable by either surgery or radiotherapy alone. This includes patients with stages IIB, IIIA, IIIB or IVA and stages IB or IIA who in addition have one of the following risk factors:

  * Primary tumor > 6 cm
  * Positive pelvic and/or para-aortic lymph nodes (resected or unresected)
  * Positive surgical margins
  * Depth of invasion greater than 50 % and positive capillary-lymphatic space involvement
  * Eligible cell types include squamous, adenosquamous and adenocarcinoma of the cervix
* Patients may have measurable disease (defined as lesions which can be measured in at least two (2) dimensions by physical examination or any medical imaging technique). Inability to measure disease will not constitute exclusion criteria.
* Patients with GOG performance status of 0, 1, or 2.
* Patients will have recovered from the effects of recent surgery and should be free of clinically significant infection.
* Patients must have adequate:

  * Bone marrow function: WBC greater than or equal to 3,000 cells/mm3, platelet count greater than or equal to 100,000 cells/mm3, and granulocyte count greater than or equal to 1,500 cells/mm3.
  * Renal function: Creatinine less than or equal to 2.0 mg/dl.
  * Hepatic function: Bilirubin less than or equal to 1.5 x institutional normal, SGOT and alkaline phosphatase less than or equal to 3 x institutional normal.
* Patients must have signed an approved informed consent.
* Patients have met the pre-entry requirements specified in Section 7.0

Exclusion Criteria:

* Patients with GOG performance of 3 or 4.
* Patients with another malignancy, prior or concomitant, other than skin (excluding melanoma).
* Patients with septicemia, severe infection, gastrointestinal bleeding, or intestinal obstruction.
* Patients with anatomic abnormalities requiring modification of radiation fields (pelvic kidney, renal transplant, etc.).
* Patient with recurrent cervical cancer
* Patients who have received prior pelvic radiation
* Pregnant women and women of childbearing potential not using an effective form of contraception.
* History of thrombus (10/28/02)
* History of unstable angina or MI within the past six months. Patients with evidence of abnormal cardiac conduction (e.g. bundle branch block, heart block) are eligible if their disease has been stable for the past six months. (10/28/02)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2002-03; Primary Completion 2004-06 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
disease progression | disease progress or complete remission

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Smith, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States